CLINICAL TRIAL: NCT05455125
Title: A Cardiac Sub-Study of the MRC National Survey of Health and Development (NSHD)
Brief Title: MultiMorbidity Life-Course Approach To Myocardial Health -A Cardiac Sub-Study of the MRC National Survey of Health and Development (NSHD)
Acronym: MyoFit46
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 123172
Record Dates: First submitted 2022-02-16; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Frailty; Cardiovascular Diseases
MeSH Terms: conditions — Frailty; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CMR CGI — High resolution ECGI plus advanced CMR

SUMMARY:
Background The life course accumulation of overt and subclinical myocardial dysfunction contributes to older age mortality, frailty, disability and loss of independence. The Medical Research Council National Survey of Health and Development (NSHD) is the world's longest running continued surveillance birth cohort providing a unique opportunity to understand life course determinants of myocardial dysfunction as part of MyoFit46-the cardiac sub-study of the NSHD.

Methods and expected results The investigators aim to recruit 550 NSHD participants of approximately 75 years+ to undertake high-density surface electrocardiographic imaging (ECGI) and stress perfusion cardiovascular magnetic resonance (CMR). Through comprehensive myocardial tissue characterization and 4-dimensional flow the investigators hope to better understand the burden of clinical and subclinical cardiovascular disease. Supercomputers will be used to combine the multi-scale ECGI and CMR datasets per participant. Rarely available, prospectively collected whole-of-life data on exposures, traditional risk factors and multimorbidity will be studied to identify risk trajectories, critical change periods, mediators and cumulative impacts on the myocardium.

Conclusion By combining well curated, prospectively acquired longitudinal data of the NSHD with novel CMR-ECGI data and sharing these results and associated pipelines with the CMR community, MyoFit46 seeks to transform our understanding of how early, mid and later-life risk factor trajectories interact to determine the state of cardiovascular health in older age.

ELIGIBILITY:
Inclusion Criteria:

* NSHD study member.
* Who is still alive and agreed to take part in the study.

Exclusion Criteria:

* Pacemaker.
* Implantable cardio defibrillator.
* Atrial fibrillation.
* Complete heart block.
* Severe asthma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NSHD cohort
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
CMR phenotype - T1 | Through study completion, an average of 4 years.
  This will be assessed through a 45 minute cardiac MRI scan with perfusion.
CMR phenotype - T2 | Through study completion, an average of 4 years.
  This will be assessed through a 45 minute cardiac MRI scan with perfusion.
CMR phenotype - Myocardial blood flow | Through study completion, an average of 4 years.
  This will be assessed through a 45 minute cardiac MRI scan with perfusion.
CMR phenotype - Aortic blood flow | Through study completion, an average of 4 years.
  This will be assessed through a 45 minute cardiac MRI scan with perfusion.

CONTACTS AND LOCATIONS:
Locations (1):
- UCL Bloomsbury Centre for Clinical Phenotyping, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Non-identifiable data sharing to external collaborators. Additional data sharing available within UCL TRE.

REFERENCES:
- [Derived] Topriceanu CC, Webber M, Shiwani H, Chan F, Martin E, Falconer D, Stanley MA, Bennett J, Gonzalez-Martin P, Shah H, De S, Wong A, Pierce I, Davies RH, Lambiase PD, Chaturvedi N, Kellman P, Hardy R, Moon JC, Hughes AD, Captur G. Higher Life-Course Blood Pressure Associates With Reduced Myocardial Perfusion in Older Age: Insights From MyoFit46. Circ Cardiovasc Imaging. 2025 Nov 8:e019105. doi: 10.1161/CIRCIMAGING.125.019105. Online ahead of print. PMID 41404671
- [Derived] Webber M, Joy G, Bennett J, Chan F, Falconer D, Shiwani H, Davies RH, Krausz G, Tanackovic S, Guger C, Gonzalez P, Martin E, Wong A, Rapala A, Direk K, Kellman P, Pierce I, Rudy Y, Vijayakumar R, Chaturvedi N, Hughes AD, Moon JC, Lambiase PD, Tao X, Koncar V, Orini M, Captur G. Technical development and feasibility of a reusable vest to integrate cardiovascular magnetic resonance with electrocardiographic imaging. J Cardiovasc Magn Reson. 2023 Dec 4;25(1):73. doi: 10.1186/s12968-023-00980-7. PMID 38044439